CLINICAL TRIAL: NCT04303130
Title: Camrelizumab (SHR-1210) Combined With Endostar for First-line Treatment in Subjects With Advanced Squamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: Camrelizumab Combined With Endostar for First-line Treatment in Subjects With Advanced Squamous NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking University First Hospital (Other); Peking University Third Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Chinese PLA General Hospital (Other); Peking Union Medical College Hospital (Other); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Fang, Director,Head of thoracic oncology, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR1210-CHEMO-BZ-201909
Record Dates: First submitted 2020-02-21; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab (SHR-1210) Combined With Endostar (Experimental): Carelizumab: PD-1 antibody SHR-1210: SHR-1210 is administered by intravenous infusion, a fixed dose of 200 mg, and intravenous infusion over 30 minutes 20 minutes, not longer than 60 minutes), once every 3 weeks, continued medication until the disease progresses intolerable toxicity and receive immunotherapy for a maximum of 2 years (35 cycles); Endo: once a day, 7.5 mg / m2 intravenous infusion, continuous administration for 14 days, rest for a week (or the corresponding dose using a micro-micropump), continued medication until disease progression toxicity intolerance.
  The combination regimen is a medication cycle every three weeks (21 days).
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Carelizumab: PD-1 antibody SHR-1210: SHR-1210 is administered by intravenous infusion, a fixed dose of 200 mg, and intravenous infusion over 30 minutes (the overall infusion time including the flushing time is not shorter than 20 minutes, not longer than 60 minutes), once every 3 weeks, continued medication until the disease progresses intolerable toxicity and receive immunotherapy for a maximum of 2 years (35 cycles); Endo: once a day, 7.5 mg / m2 intravenous infusion, continuous administration for 14 days, rest for a week (or the corresponding dose using a micro-micropump), continued medication until disease progression toxicity intolerance.
  The combination regimen is a medication cycle every three weeks (21 days).
  Other Names: Endostar

SUMMARY:
This study is a single-arm, prospective, multi-center clinical trial. designed to evaluate patients with stage IV inability to receive or refuse chemotherapy.Efficacy and safety of first-line treatment with Camrelizumab and Endo in advanced lung squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Subjects >/= 18 years of age at the time of Informed Consent.
2. Subjects with histopathological diagnosis of squamous non-small cell lung cancer (SqNSCLC) have a histologically or cytologically confirmed stage IV (American Joint Committee on Cancer [AJCC] 8th edition) , and the stage IIIB/IIIC SqNSCLC that is unresectable and not fit for radical concurrent chemoradiotherapy.
3. .No prior systemic treatment. Subjects who have received prior neo-adjuvant, adjuvant chemotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment free interval of at least 6 months from randomization since the last chemotherapy cycle.
4. Life expectancy of at least three months.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Subjects enrolled must have measurable lesion(s) according to the RECIST 1.1 standard (the CT scan length of the tumor lesion > 10 mm, the short diameter of CT scan of the lymph node lesions > 15 mm).
7. The main organ function is normal. All baseline laboratory requirements will be assessed and should be obtained within -14 days of randomization. Screening laboratory values must meet the following criteria.

   1. Hemoglobin ≥ 9.0 g/dL (90 g/L)
   2. Absolute neutrophil count ≥ 2× 109/L
   3. Platelets ≥ 100× 109/L
   4. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN)
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal(ULN); alkaline phosphatase ≤ 5 × ULN
   6. Serum creatinine ≤ 1× ULN or creatinine clearance > 60 mL/minute (using Cockcroft/Gault formula)
8. Subject dosen't have unhealed wounds before enrollment.
9. Female participants of childbearing potential must have a negative serum pregnancy test within -7 days of randomization and must be willing to use very efficient barrier methods of contraception or a barrier method plus a hormonal method starting with the screening visit through 60 days (about 5 drug half-life + menstrual cycle) after the last dose of SHR-1210. Male participants with a female partner(s) of child-bearing potential must be willing to use very efficient barriermethods of contraception from screening through 120 days (about 5 drug half-life + sperm depletion cycle) after the last dose of SHR-1210.
10. Subjects should be voluntarily participate in clinical studies and informed consent should be signed.

Exclusion Criteria

1. Active central nervous system (CNS) metastasis and/or cancerous meningitis. Patients with treated brain metastases who were clinically stable for at least 2 weeks and have no new or advanced brain metastases may be enrolled. Patients with known untreated, asymptomatic brain metastases can be enrolled provided cerebral imaging assessment be regularly performed.
2. Subjects used immunosuppressive drugs excluding nasal spray and inhaled corticosteroids or systemic steroids at physiological doses(prednisolone≤10 mg/day or other corticosteroids of the same pharmacophysiological dose) within 14 days before the first dose.
3. Subjects with grade II or above myocardial ischemia or myocardial infarction and poorly controlled arrhythmias (QTc interval > 450 ms for males and QTc interval > 470 ms for females). Subjects with grade III-IV cardiac insufficiency or with left ventricular ejection fraction (LVEF) less than 50% had myocardial infarction within 6 months before admission according to NYHA criteria. Subjects with uncontrolled hypertension.
4. Participants who had any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis , Hyperthyroidism, decreased thyroid function).
5. subjects with childhood asthma has completely resolved, adults can be included without any intervention; subjects with bronchodilators for medical intervention can not be included .
6. Participants who had abnormal blood coagulation (INR>1.5 or PT> ULN+4s, and or APTT > 1.5 ULN), bleeding tendency or receiving thrombolytic or anticoagulation；
7. Urine routine indicates urinary protein ≥ ++, or confirms that 24-hour urine protein is ≥1.0 g；
8. Patients with non-healing wound, non-healing ulcer, or non-healing bone fracture;
9. The patient has severe infection within 4 weeks before first administration（such as the need for intravenous antibiotics, antifungals or antivirals) and unexplained fever within 7 days before administration, ≥38.5 °C
10. There was significant coughing blood and significant clinically significant bleeding symptoms or a clear tendency to hemorrhage in the first 2 months before enrollment (such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ and above at baseline, or suffering from vasculitis, etc.).
11. Serious Arterial / venous thrombosis events, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism, within 12 months before enrollment.
12. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection. (HBV: HBsAg positive and HBV DNA ≥ 500 IU/mL ; HVC: HCV RNA positive and abnormal liver function). And subjects with active tuberculosis.
13. History of severe hypersensitivity reactions to any component contained in Endostar or antibody preparation of Camrelizumab. And known to have severe allergic reactions to infusion reactions.
14. Any known mental illness or substance abuse that may have an impact on compliance with the test requirements;
15. There are other factors lead to patients can not participate in this clinical study by the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free survival) | 1 Year
  From the date Into this study (signed ICF) to tumor progression or death for any
One year survival rate | 1 Year

SECONDARY OUTCOMES:
ORR (Objective control rate) | From the date Into this study (signed ICF) to tumor progression，assessed up to 36 months.
  The rate of CR and PR
DCR (Disease control rate) | From the date Into this study (signed ICF) to tumor progression，assessed up to 36 months.
  the rate of CR, PR plus SD
DOR(Duration of response） | From the date Into this study (signed ICF) to tumor progression，assessed up to 36 months.
  Cr or PR to the first assessment of PD or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jian Fang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China